CLINICAL TRIAL: NCT04550481
Title: Role of Lisinopril in Preventing The Progression of Non-Alcoholic Fatty Liver Disease (NAFLD): Relief-NAFLD
Brief Title: Role of Lisinopril in Preventing the Progression of Non-Alcoholic Fatty Liver Disease, RELIEF-NAFLD Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2020-06905; NCI-2020-06905 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI20-01-03 (Other: Northwestern University); NWU20-01-03 (Other: DCP); P30CA060553 (NIH); UG1CA242643 (NIH)
Record Dates: First submitted 2020-09-15; First posted 2020-09-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Non-alcoholic Fatty Liver Disease | interventions — Specimen Handling; Lisinopril; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (lisinopril) (Experimental): Patients receive lisinopril PO QD for 24 weeks in absence of unacceptable toxicity. Patients undergo transient elastography during screening and on study. Patients also undergo blood sample collection on study and may undergo a PDFF MRI and MRE on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Lisinopril; Procedure: Liver Ultrasonographic Elastography; Procedure: Magnetic Resonance Elastography; Procedure: Magnetic Resonance Imaging; Procedure: Proton Density Fat Fraction; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Lisinopril — Given PO
  Other Names: N2-[(1S)-1-Carboxy-3-phenylpropyl]-L-lysyl-L-proline, Dihydrate; Prinivil; Zestril
Procedure: Liver Ultrasonographic Elastography — Undergo transient elastography
  Other Names: Fibroscan; TE; Transient Elastography; VCTE; Vibration-Controlled Transient Elastrography
Procedure: Magnetic Resonance Elastography — Undergo PDFF MRE
  Other Names: MRE
Procedure: Magnetic Resonance Imaging — Undergo PDFF MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Proton Density Fat Fraction — Undergo PDFF MRI/MRE
  Other Names: Fat Fraction by Proton Density; PDFF
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial investigates how well lisinopril may work in preventing the progression of non-alcoholic fatty liver disease (NAFLD). NAFLD is a condition where there is an accumulation of fatty cells in the liver. NAFLD increases a person's risk of developing liver cancer. Liver fibrosis is the common finding of chronic liver diseases leading to reduced liver function. Lisinopril is a medication that is commonly used to treat high blood pressure. Lisinopril may help to decrease liver fibrosis. The purpose of this trial is to find out what effect, if any, lisinopril has on a patient's risk of developing liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if NAFLD patients with advanced fibrosis will demonstrate a change in PRO-C3, a marker of liver fibrosis, following 24 weeks of treatment with lisinopril.

SECONDARY OBJECTIVES:

I. Noninvasive measures of fibrosis and steatosis:

Ia. Change from baseline in PC3X (cross-linked multimeric PRO-C3);

Ib. Change from baseline in steatosis, as measured by controlled attenuation parameter (CAP) or liver ultra-sound attenuation (LiSA), determined with transient elastography:

Ic. Change from baseline in liver stiffness as measured with magnetic resonance elastography (MRE); Id. Change from baseline in liver stiffness as measured with transient elastography; Ie. Changes from baseline in Fibrosis-4 score (FIB-4) and NAFLD fibrosis score (NFS); If. Change in inflammatory markers (caspase cleaved cytokeratin 18 [CK-18], NF-kappaB, TGF-beta, TNF-alpha, IL6 and IL8).

OUTLINE:

Patients receive lisinopril orally (PO) once daily (QD) for 24 weeks in absence of unacceptable toxicity. Patients undergo transient elastography during screening and on study. Patients also undergo blood sample collection on study and may undergo a proton density fat fraction (PDFF) magnetic resonance imaging (MRI) and MRE on study.

Patients are followed up at 32 weeks after the start of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects >= 18 years of age
* Clinical diagnosis of nonalcoholic steatohepatitis (NASH) assessed by the presence of body imaging criteria (ultrasound, computed tomography [CT], or magnetic resonance imaging [MRI]), or liver biopsy up to six months prior to enrollment without suspicious nodules or cancer
* Screening transient elastography liver stiffness >= 12 kPa (which correlates with F3 fibrosis and more) and < 25 kPa. Historic transient elastography within 0-4 weeks prior to the date of the screening visit is acceptable. Patients with liver stiffness >= 10 and < 12 kPA with clinical evidence of cirrhosis based on any of the following criteria would also be eligible.

  * Imaging diagnosis of nodular liver with splenomegaly or recanalized umbilical vein
  * MRE >= 5 kPa
  * Fibrosis (FIB)-4 > 2.67 or platelet count < 150,000 mL
  * Liver biopsy < 5 years with meta-analysis of histological data in viral hepatitis (METAVIR) stage 4 or Ishak stage 5-6
* Controlled attenuation parameter score or liver steatosis analysis (LiSA) of >= 260 dB/m and any single component of metabolic syndrome (ATP3 criteria) or historic liver biopsy within 0 - 6 months prior to the date of the screening visit consistent with nonalcoholic steatohepatitis (NASH) (defined as the presence of steatosis, inflammation, and ballooning), with stage 3-4 fibrosis according to the NASH Clinical Research Network classification (or equivalent)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 75,000/microliter
* Total bilirubin within normal institutional limits unless the patient has Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 8 x institutional upper limit of institutional limits
* Glomerular filtration rate > 30 ml/min
* International normalized ratio (INR) =< 1.3 unless the patient is on a therapeutic medication
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* The effects of lisinopril has been shown to be teratogenic in animal models. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document. If a participant has impaired decision-making capacity (IDMC), their legal representative may replace them in this process
* Systolic blood pressure >= 90 and =< 160 mm/Hg. Diastolic blood pressure >= 60 and =< 110 mm/Hg

Exclusion Criteria:

* Prior or current use of an angiotensin converting enzyme inhibitor (ACEi) or angiotensin II receptor antagonist (ARB) within 0-24 weeks prior to enrollment
* Glomerular filtration rate =< 30 ml/min (for both male and female participants)
* History of decompensated liver disease, including ascites, hepatic encephalopathy, or high-risk variceal bleeding

  * NOTE: Trace ascites documented by radiology is permitted
* History of other causes of liver disease, including but not limited to alcoholic liver disease, hepatitis B, hepatitis C, autoimmune disorders (primary biliary cholangitis, primary sclerosing cholangitis, or autoimmune hepatitis), drug-induced hepatotoxicity, Wilson's disease, iron overload, or alpha-1-antitryspin deficiency
* History of liver transplantation
* History of hepatocellular carcinoma (HCC) diagnosis
* History of weight reduction surgery in the past 2 years or planned during the study
* Within 6 months prior to the date of the screening visit, there must be no history of the following cardiac events: unstable angina; myocardial infarction, coronary artery bypass surgery or coronary angioplasty; transient ischemic attack or cerebrovascular accident; emergency room visit or hospitalization for confirmed cardiovascular disease
* Participants taking vitamin E >= 800 IU/day must be on a stable dose, defined as no changes in prescribed dose, new vitamin E-containing medications, or discontinuation for at least 180 days prior to the date of the screening visit and throughout study participation
* Participants taking anti-diabetic medications must be on a stable dose for at least 90 days prior to the date of the screening visit and in the period between the date of the screening visit and enrollment
* Current alcohol consumption > 21 oz/week for males or > 14 oz/week for females (1 oz/30 mL of alcohol is present in one 12 oz/360 mL beer, 4 oz/120 mL glass of wine, and a 1oz/30 mL measure of 40 proof [20%] alcohol)
* Participants may not be receiving any other investigational agents, at the time of the screening visit, or in the prior 30 days, or within 5 half-lives of the prior investigational agent (whichever is longer)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lisinopril
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* History of human immunodeficiency virus (HIV) infection. HIV patients may develop fatty liver as well as advanced fibrosis due to many causes including metabolic syndrome, hyperuricemia, HIV-related lipodystrophy, genetic polymorphisms, medications, and HIV itself. As the natural history of fatty liver in this population is largely unknown, these patients will be excluded from this study
* Women who are pregnant or breastfeeding. Pregnant women are excluded from this study because lisinopril is an ACE Inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with lisinopril. Breastfeeding should be discontinued if the mother is treated with lisinopril
* Systolic blood pressure >= 161 mm/Hg. Diastolic blood pressure >= 111 mm/Hg
* Participants taking lithium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in PRO-C3 values | Baseline to 24 weeks
  Descriptive statistics will be used to summarize changes and values at each time point. The primary analysis will be performed using a paired t-test to compare the pre- to post-treatment changes in PRO-C3 levels. PRO-C3 levels will be log-transformed to satisfy the normality assumption. If log-transformation does not satisfy the normality assumption, a signed rank test will be used.

SECONDARY OUTCOMES:
Change in PC3X (cross-linked multimeric PRO-C3) | Baseline to 24 weeks
Change in steatosis | Baseline to 24 weeks
  Measured by controlled attenuation parameter or liver steatosis analysis, determined with transient elastography. Changes in categorical variables will be analyzed using the Stuart-Maxwell test of marginal homogeneity. Linear regression models will be used to identify baseline characteristics that are associated with biomarker changes. Model selection will be conducted according to the purposeful model selection approach (REF) to a parsimonious set of predictors. Model fit will be assessed using standard regression diagnostics. Changes in categorical outcomes from pre- to post-treatment will also be categorized as improvement vs. no improvement (i.e. no change or worsening in steatosis grade), and logistic regression models will be used to examine association with baseline characteristics.
Change liver stiffness | Baseline to 24 weeks
  Measured with magnetic resonance elastography. Changes in categorical variables will be analyzed using the Stuart-Maxwell test of marginal homogeneity. Linear regression models will be used to identify baseline that are associated with biomarker changes. Model selection will be conducted according to the purposeful model selection approach (REF) to a parsimonious set of predictors. Model fit will be assessed using standard regression diagnostics. Changes in categorical outcomes from pre- to post-treatment will also be categorized as improvement vs. no improvement (i.e. no change or worsening in steatosis grade), and logistic regression models will be used to examine association with baseline characteristics.
Change liver stiffness | Baseline to 24 weeks
  Measured with transient elastography. Changes in categorical variables will be analyzed using the Stuart-Maxwell test of marginal homogeneity. Linear regression models will be used to identify baseline characteristics that are associated with biomarker changes. Model selection will be conducted according to the purposeful model selection approach (REF) to a parsimonious set of predictors. Model fit will be assessed using standard regression diagnostics. Changes in categorical outcomes from pre- to post-treatment will also be categorized as improvement vs. no improvement (i.e. no change or worsening in steatosis grade), and logistic regression models will be used to examine association with baseline characteristics.
Change in non-alcoholic fatty liver disease (NAFLD) fibrosis score (NFS) | Baseline to 24 weeks
  Changes in categorical variables will be analyzed using the Stuart-Maxwell test of marginal homogeneity. Linear regression models will be used to identify baseline characteristics that are associated with biomarker changes. Model selection will be conducted according to the purposeful model selection approach (REF) to a parsimonious set of predictors. Model fit will be assessed using standard regression diagnostics. Changes in categorical outcomes from pre- to post-treatment will also be categorized as improvement vs. no improvement (i.e. no change or worsening in steatosis grade), and logistic regression models will be used to examine association with baseline characteristics.
Change in Fibrosis-4 score | Baseline to 24 weeks
  Changes in categorical variables will be analyzed using the Stuart-Maxwell test of marginal homogeneity. Linear regression models will be used to identify baseline characteristics that are associated with biomarker changes. Model selection will be conducted according to the purposeful model selection approach (REF) to a parsimonious set of predictors. Model fit will be assessed using standard regression diagnostics. Changes in categorical outcomes from pre- to post-treatment will also be categorized as improvement vs. no improvement (i.e. no change or worsening in steatosis grade), and logistic regression models will be used to examine association with baseline characteristics.
Change in inflammatory markers (caspase cleaved cytokeratin 18, NF-kappaB, TGF-beta, TNF-alpha, IL6 and IL8) | Baseline to 24 weeks
  Descriptive statistics, including means, 95% confidence intervals, or median and inter-quartile range, will be used to summarize changes as well as biomarker values at each time point. To determine whether changes in these biomarkers occurred following treatment, paired t-test will be used as described for the analysis of the primary endpoint. Biomarker values may be transformed to satisfy the normality assumption. If no suitable transformation can be found, a signed rank test will be used. For the analysis of inflammatory biomarkers, tests will be adjusted for multiple comparisons to control the false discovery rate using the method of Romano.

OTHER OUTCOMES:
Change in steatosis | Baseline to 24 weeks
  Measured by magnetic resonance imaging-proton density fat fraction. Changes in categorical variables will be analyzed using the Stuart-Maxwell test of marginal homogeneity. Linear regression models will be used to identify baseline characteristics that are associated with biomarker changes. Model selection will be conducted according to the purposeful model selection approach (REF) to a parsimonious set of predictors. Model fit will be assessed using standard regression diagnostics. Changes in categorical outcomes from pre- to post-treatment will also be categorized as improvement versus (vs.) no improvement (i.e. no change or worsening in steatosis grade), and logistic regression models will be used to examine association with baseline characteristics.
Change in markers of liver injury and function: alanine aminotransferase, aspartate aminotransferase, bilirubin, and alkaline phosphatase | Baseline to 24 weeks
Change in homeostatic assessment of glycosylated hemoglobin | Baseline to 24 weeks
Change in serum lipid profiles | Baseline to 24 weeks
Change in systolic and diastolic blood pressure | Baseline to 24 weeks
Changes in microbiome and metabolomics and genomics | Baseline to 24 weeks
  Collect urine, stool, serum/plasma, and genomic deoxyribonucleic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Ju Dong Yang, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm